CLINICAL TRIAL: NCT05155813
Title: Prevalence of Sleep Apnea Among Consecutive Patients With Atrial Fibrillation.
Brief Title: Prevalence of Sleep Apnea and Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Itamar-Medical, Israel (Industry)
Responsible Party: Principal Investigator, Sogol Javaheri, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2021P002370
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Sleep Apnea; Atrial Fibrillation
Keywords: sleep apnea; atrial fibrillation
MeSH Terms: conditions — Sleep Apnea Syndromes; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: WatchPAT — FDA-approved portable home sleep testing device worn on the wrist.

SUMMARY:
The investigators will screen consecutive patients presenting to the atrial fibrillation clinic for sleep apnea using a FDA-approved home sleep testing device, WatchPAT to determine prevalence of sleep apnea in a clinic-based sample.

DETAILED DESCRIPTION:
The investigators will determine the prevalence of sleep apnea among consecutive patients with atrial fibrillation (AF) regardless of symptoms and determine the predictive value of screening tools for sleep apnea in this population. The primary outcome will be the prevalence of sleep apnea among all-comers with AF. Three secondary outcomes will be evaluated in the study. Investigators will determine the efficiency and time-to-diagnosis of sleep apnea using a FDA approved home sleep testing device (i.e. WatchPAT). These analyses will be compared to published studies performed using a traditional home sleep study test (which historically takes approximately 8-10 weeks). There will be no collection of data from a non-intervention group in our study. Second, investigtaors will calculate the predictive value of traditional clinical screening tools in an AF population using the STOP-BANG questionnaire and Epworth Sleepiness Scale. Third, investigators will identify potential risk factors for AF in patients with sleep apnea using a logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AF confirmed on any electrocardiographic recording
* Age greater than or equal to 18
* Ability to read and understand consent form, complete questionnaires, and provide informed consent

Exclusion Criteria:

* Prior diagnosis of sleep disordered breathing or negative testing within the past 2 years without significant change in weight or clinical symptoms of sleep apnea
* History of Raynaud

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are referred to the Atrial Fibrillation Center of Excellence by their primary care provider or primary cardiologist will be screened by eligibility by study staff during their first clinic visit (in-person or virtually).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sleep apnea | 2 year study
  Prevalence of sleep apnea among patients with atrial fibrillation

SECONDARY OUTCOMES:
Time to diagnosis | 2 years
  We will determine the efficiency and time-to-diagnosis of sleep apnea using a FDA approved home sleep testing device (i.e. WatchPAT)
Predictive value of typical screening tools | 2 years
  We calculate the predictive value of traditional clinical screening tools in an AF population using the STOP-BANG questionnaire and Epworth Sleepiness Scale
Quality of life | 2 years
  We will compare quality of life using the MAFSI in atrial fibrillation patients with and without sleep apnea.
Risk factors | 2 years
  We will identify potential risk factors for AF in patients with sleep apnea using a logistic regression model

OTHER OUTCOMES:
Autonomic index | 2 years
  Compare autonomic index in patients with AF who have sleep apnea versus those without sleep apnea
Insomnia Severity Index | 2 years
  Assess prevalence of insomnia among consecutive patients with atrial fibrillation

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mills EW, Cassidy M, Sofer T, Tadros T, Zei P, Sauer W, Romero J, Martin D, Antman EM, Javaheri S. Evaluation of obstructive sleep apnea among consecutive patients with all patterns of atrial fibrillation using WatchPAT home sleep testing. Am Heart J. 2023 Jul;261:95-103. doi: 10.1016/j.ahj.2023.03.014. Epub 2023 Apr 3. PMID 37019195